CLINICAL TRIAL: NCT02413931
Title: Nosocomial Transmission of Multidrug-resistant Tuberculosis at the Marius Nasta Institute in Bucharest, Romania
Brief Title: Nosocomial Transmission of MDR-TB in Bucharest, Romania
Status: Completed | Type: Observational
Sponsor: Research Center Borstel (Other)
Collaborators: "Marius Nasta" Pulmonology Institute (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Christoph Lange, Chief investigator, Research Center Borstel
Other Study IDs: RCBorstel_MNI_001
Record Dates: First submitted 2015-03-17; First posted 2015-04-10 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Tuberculosis, Multidrug-resistant
Keywords: tuberculosis; MDR-TB
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum, blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with MDR-TB: Patients with multidrug-resistant tuberculosis admitted for treatment at the Marius Nasta Institute will be included
  Interventions: Other: Routine management practices applied

INTERVENTIONS:
Other: Routine management practices applied — all patients will be treated according to routine procedures, no intervention

SUMMARY:
It is a single-center, observational, prospective cohort study recruiting patients hospitalized at the multidrug-resistant tuberculosis ward at Marius Nasta Institute. This project aims to improve the individual patient management and TB treatment outcomes, especially for patients with drug-resistant TB and/or co-morbidities. The study will be conducted in a co-operation between the Marius Nasta Institute, Division of Infectious Diseases & Tropical Medicine of Klinikum of the University of Munich (KUM) and the German Center for Infection Research (DZIF).

DETAILED DESCRIPTION:
Although in Germany tuberculosis (TB) is becoming a rare disease, TB continues to represent a major cause of morbidity and mortality worldwide. According to the World Health Organization, more than 10 million TB cases were registered worldwide leading to 1.8 million deaths. In the absence of a vaccine that is more effective to prevent TB than the M. bovis Bacille Calmette Guérin vaccine, TB prevention will rely on early case detection and preventive therapies for individuals who are latently infected with M. tuberculosis. Treatment of active TB requires taking a combination of anti-mycobacterial drugs for a very long time to achieve relapse-free cure. Current international guidelines recommend treatment for pan-drug susceptible pulmonary TB for 6 months, more importantly, a total of 20 months is recommended for treatment of patients with M/XDR-TB. These general recommendations are not applicable to the majority of affected patients. A substantial proportion of patients with TB will achieve relapse-free cure with shorter durations of anti-mycobacterial treatments. However, biomarkers that guide clinicians to decide on the individual duration of TB therapy are lacking. Optimal duration of TB treatment depends on a variety of variables, such as the extent of disease, the immune-status of the host, co-morbidities/infections, drug-resistance and virulence of the causative bacilli, and availability of anti-mycobacterial drugs. For many patients, especially those affected by M/XDR-TB, the long duration of therapy is related to substantial morbidity and loss of quality of life due to adverse events of the treatment.

This project has the goal to further the development of the previously established good clinical practice (GCP)-conform clinical study site at the Marius Nasta Institute (MNI) in Bucharest, Romania. The Eastern European Study Site will represent and important partner and support the conduction of a number of studies within other work packages as well as continue the enrollment of patients with multidrug-resistant (MDR) and extensively drug-resistant (XDR) tuberculosis (TB) started earlier. The characteristics of patients with M/XDR-TB and co-morbidities of patients with TB will be recorded and their influence on patient outcome will be analyzed. In this setting, biomarkers that could help individualize the duration of anti-tuberculosis therapy and that could offer an early prediction of treatment outcome will be validated. The study site could also provide a platform for the conduction of studies aimed at developing and standardizing a system of drug-level monitoring (therapeutic drug monitoring) for TB. The project will therefore support studies with the goal of individualizing therapy for TB and represent a valuable international DZIF-partner in a medium-TB-incidence setting. Within this project, the partnership with the good clinical practice (GCP)-conform Eastern European Study Site at the Marius Nasta Institute MNI) in Bucharest, Romania will be continued. The MNI is the country-wide referral center for the treatment of M/XDR-TB in Romania and hosts the Romanian Reference Laboratory for Mycobacteria.

This project aims to improve the individual patient management and TB treatment outcomes, especially for patients with drug-resistant TB and/or co-morbidities. This will be achieved by:

* Identify characteristics of patients with M/XDR-TB from the MNI. This could potentially lead to the identification of risk factors associated with drug-resistant TB in Romania, predictors of an unsuccessful treatment outcome, as well as record management practices of patients with M/XDR-TB.
* Analysis of transmission routes and molecular drug-resistance profiles of M. tuberculosis strains isolated from M/XDR to differentiate between nosocomial and community acquired infections.
* Further development of the already established GCP-conform Eastern European Study Site.
* Identification and validation of bio-signatures to allow treatment outcome prediction and evaluation of markers that will eventually guide clinicians for decisions on the durations of therapy
* Evaluation of co-morbidities/infections and inflammation status on TB treatment outcome
* Evaluation of cardio-pulmonary TB-outcome (e.g. lung function) as a clinical marker to describe treatment success/treatment outcome
* Evaluation of neutrophils as targets for host-directed therapies and neutrophil signatures from bronchial secretions for point-of-care diagnosis
* Evaluation of lipids as targets for host-directed therapies and lipid signatures from bronchial secretions for point-of-care diagnosis
* Establishment and evaluation of therapeutic drug monitoring techniques for anti-mycobacterial therapy regimens

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with confirmed pulmonary MDR-TB
2. Subject able and willing to give informed consent

Exclusion Criteria:

1. physical or mental inability preventing study participation at the discretion of the investigator
2. member of a vulnerable or special population (prisoner, soldier, mentally ill, under guardianship,
3. age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with microbiologically confirmed pulmonary MDR-TB admitted to the MDR-TB ward of the Marius Nasta Instiute
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-05; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with nosocomially transmitted MDR-TB | until the end of treatment - ca. 20 months after enrolment

SECONDARY OUTCOMES:
Concordance between phenotypic drug susceptibility testing and detected resistance mutations | until the end of treatment - ca. 20 months after enrolment
Proportion of patients with changes in drug susceptibility pattern during treatment | until the end of treatment - ca. 20 months after enrolment
Proportion of patients with mixed infections | until the end of treatment - ca. 20 months after enrolment
Clustering within the MDR-TB patient population | until the end of treatment - ca. 20 months after enrolment
Number of patients with different TB genotypes (e.g. Beijing, LAM, EAI, etc.) | until the end of treatment - ca. 20 months after enrolment
Proportion of patients with cardio-pulmonary impairment at different time points | until the end of treatment - ca. 48 months after enrolment
Proportion of patients with socio-economic and psychological adverse outcomes | until the end of treatment - ca. 48 months after enrolment
Proportion of patients with co-morbidities and co-infections | until the end of treatment - ca. 48 months after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Lange, MD, PhD, Principal Investigator — Research Center Borstel
Locations (1):
- Marius Nasta Pulmonology Institute, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided
this will be decided at a later time point